CLINICAL TRIAL: NCT04521855
Title: The Caregiver's Burden in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Tatiana Besse-Hammer (Other)
Responsible Party: Sponsor-Investigator, Tatiana Besse-Hammer, Head of the clinical trial unit, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Other Study IDs: CHUB-Lombardo
Record Dates: First submitted 2020-08-18; First posted 2020-08-21 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Caregivers: Caregivers (family environment or close entourage) for adults and children with cerebral palsy.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaires in French on the quality of life, the burden of caregiving and a screening for depressive symptoms, completed during specific interviews.

SUMMARY:
Cerebral palsy (CP) results from damage to the developing brain of the fetus or infant. These non-progressive lesions cause a set of permanent movement and posture disorders, responsible for activity limitations. These disorders are often accompanied by sensory, perceptual, cognitive impairments, communication and behavioral disorders, and sometimes epilepsy and/or secondary musculoskeletal problems. It is the leading cause of motor disability in childhood and affects 200 newborns per year in Belgium.

Cerebral palsy affects two to three people in every 1,000 of the world's population. The prevalence, incidence and most common causes have varied over time due to significant changes in obstetric care and pediatric care. In 75% of all cases of cerebral palsy, the lesions occurred before childbirth.

The population of adults diagnosed with cerebral palsy is increasing as the survival rate of children born with a disability increases. This population requires adapted and expert care services for the continuous monitoring and management of their condition. In addition, the development of additional health problems in adulthood increases the need for permanent access to care structures. Adults with CP have a higher rate of chronic health problems (ischemic heart disease) and a deterioration in their functional status. They would also have difficulty having a social and professional life which negatively impacts their quality of life.

A large number of adults with CP cannot access appropriate care or medico-social structures. This results in a significant involvement of caregivers (family environment or close entourage).

The role of caregiver is at the origin of a significant physical and psychological burden, whether for underage patients or adult patients. The study of this burden is well known in certain neurological pathologies (head trauma, multiple sclerosis, brain tumors). In the field of cerebral palsy, a study showed that the primary caregivers of children with CP had higher levels of psychological and physical disorders than the control group studied (caregivers of healthy children).

Currently, there are very few studies assessing the burden of caregivers of adults with cerebral palsy. The objective of this study is to analyze, through various specific questionnaires, the quality of life and the presence of depressive symptoms linked to the burden of caregivers of adults and children with cerebral palsy, taking into account socio-economic and environmental data.

ELIGIBILITY:
Inclusion Criteria:

- Healthy subjects, aged 18 to 75, caring for relatives of adults and children with cerebral palsy, with a good understanding of the French language.

Exclusion Criteria:

- Subjects under 18 or over 75, presenting a language barrier (interview guide written in French), subjects with a known history of psychiatric pathologies.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy subjects, aged 18 to 75, caring for relatives of adults and children with cerebral palsy, with a good understanding of the French language.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-10-05 (Actual); Study Completion 2022-10-05 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and depression scale (HAD) | 15 minutes
  The HAD scale is an instrument used to screen for anxiety and depressive disorders. An overall score is calculated by adding the responses to the 14 items (varies from 0 to 42) as well as two sub-scores corresponding to the two subscales (ranging from 0 to 21). The higher the scores, the more severe the symptomatology.
ISPN (Nottingham Health Profile - NHP) | 15 minutes
  The Nottingham Health Profile (NHP) is a general patient reported outcome measure which seeks to measure subjective health status. All questions have only yes/no answer options and each section score is weighted. The higher the score, the greater the number and severity of problems. The highest score in any section is 100.
Zarit scale | 15 minutes
  The Zarit scale assesses the burden felt by caregivers. The total score, which is the sum of the scores obtained for each of 22 items, varies from 0 to 88. A lower score or equal to 20 indicates little or no charge; a score between 21 and 40 indicates a light load; a score between 41 and 60 indicate a moderate load; a score above 60 indicates a severe load.
SF12 | 15 minutes
  The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is often used as a quality of life measure. A high score corresponds to a better state of health.

CONTACTS AND LOCATIONS:
Overall Officials: Costanza Lombardo, MD, Principal Investigator — CHU Brugmann
Locations (1):
- Brugmann University Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No